CLINICAL TRIAL: NCT03230916
Title: A Phase 1b, Open-label, Single-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of MK-7655A in Pediatric Subjects From Birth to Less Than 18 Years of Age With Confirmed or Suspected Gram-negative Infections
Brief Title: A Pharmacokinetics Study of MK-7655A in Pediatric Participants With Gram-negative Infections (MK-7655A-020)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7655A-020; MK-7665A-020 (Other: Merck); 2016-004328-43 (EudraCT Number)
Record Dates: First submitted 2017-07-17; First posted 2017-07-27 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Suspected or Documented Gram-negative Bacterial Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMI/REL FDC (Experimental): Imipenem/Cilastatin/Relebactam (IMI/REL) administered as a single fixed 2:1 ratio of imipenem/cilastatin to relebactam, with a maximum dose of 15 mg/kg IMI and 15 mg/kg CIL (up to 500 mg IMI and 500 mg CIL) and 7.5 mg/kg REL (up to 250 mg REL).
  Interventions: Drug: IMI/REL FDC

INTERVENTIONS:
Drug: IMI/REL FDC — IMI/REL is supplied as a single fixed dose combination (FDC) vial; which is administered at a maximum dose of 15 mg/kg IMI and 15 mg/kg CIL (up to 500 mg IMI and 500 mg CIL) and 7.5 mg/kg REL (up to 250 mg REL).
  Other Names: MK-7655A

SUMMARY:
This study aims to obtain plasma pharmacokinetic (PK) data and characterize the PK profile of imipenem (IMI), cilastatin (CIL), and relebactam (REL) following administration of a single intravenous (IV) dose of MK-7655A (a fixed ratio combination of imipenem/cilastatin/relebactam), hereafter referred to as IMI/REL.

ELIGIBILITY:
Inclusion Criteria:

* Has a parent or legally acceptable representative (LAR) who provides written informed consent for the trial on the participant's behalf.
* Aged from birth to <18 years old.
* Is hospitalized, currently receiving antibacterial treatment for confirmed or suspected Gram-negative bacterial infection, and expected to require hospitalization until at least 24 hours after completion of study drug administration.
* Is not of reproductive potential; but if of reproductive potential, agrees to avoid becoming pregnant or impregnating a partner from the time of consent through 24 hours after completion of study drug administration.
* Has clinically stable renal function at the time of screening that is judged to be within acceptable ranges.
* Has sufficient intravascular access to receive study drug through an existing peripheral or central line.

Exclusion Criteria:

* Has a personal history of hypersensitivity to imipenem/cilastatin (IMI) or to any of the following: any carbapenem, cephalosporin, penicillin, or other β-lactam agent; or other β-lactamase inhibitors (BLIs) e.g. tazobactam, sulbactam, clavulanic acid, avibactam.
* Female is currently pregnant or breast feeding or has a positive serum β-human chorionic gonadotropin (β-hCG) pregnancy test.
* Has a history of a seizure disorder requiring ongoing treatment with anti-convulsive therapy or prior treatment with anti-convulsive therapy within the last 3 years.
* Has used or plans to use valproic acid or divalproex sodium within 2 weeks prior to screening or at any point between screening and 24 hours after the completion of study drug infusion.
* Has received treatment or plans to receive treatment with any carbapenem antibiotic within 48 hours prior to initiation of study drug infusion or at any point between administration of study drug and the last PK sample collection.
* Has used or plans to use any of the following medications, which are organic anion transporter (OAT) 1 or OAT3 inhibitors, within 1 week prior to screening or at any point between screening and the last PK sample collection: cimetidine, probenecid, indomethacin, mefenamic acid, furosemide or other loop diuretics (eg, bumetanide, torsemide, ethacrynic acid), angiotensin receptor blockers (eg, valsartan), and ketorolac.
* Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 30 days prior to screening.
* Has enrolled previously in the current trial and been discontinued, or has received REL for any other reason.
* Has a current diagnosis of cystic fibrosis, meningitis, or severe sepsis.
* Is expected to survive less than 72 hours after completion of study drug administration.
* Has a history of clinically significant renal, hepatic, or hemodynamic instability.
* Plans to use cardiopulmonary bypass, extracorporeal membrane oxygenation, hemodialysis, or peritoneal dialysis during the study.
* For participants that are 2 to 17 years of age only: weighs outside of the 5th to 95th percentile based on age.
* Is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence.
* Has a planned blood transfusion within 24 hours of study drug administration or expected before the end of the PK sampling.
* Has had significant blood loss (≥5% of total blood volume) within 4 weeks before the screening visit.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (33):
- United States (8):
  - Arkansas Children's Hospital ( Site 1311), Little Rock, Arkansas
  - Children's Hospital of Orange County ( Site 1301), Orange, California
  - Rady Children's Hospital-San Diego ( Site 1305), San Diego, California
  - Our Lady of the Lake Hospital ( Site 1304), Baton Rouge, Louisiana
  - St. Louis Children's Hospital ( Site 1322), St Louis, Missouri
  - Duke University Medical Center ( Site 1317), Durham, North Carolina
  - The Children's Hospital of Philadelphia ( Site 1318), Philadelphia, Pennsylvania
  - Seattle Childrens Hospital ( Site 1321), Seattle, Washington
- Bulgaria (5):
  - MHAT Pazardjik AD ( Site 0208), Pazardzhik, Pazardzhik
  - UMHAT Deva Maria. EOOD ( Site 0209), Burgas
  - UMHAT Dr. Georgi Stranski EAD ( Site 0211), Pleven
  - UMHAT Kanev AD ( Site 0203), Rousse
  - UMHAT Kanev AD ( Site 0212), Rousse
- Colombia (3):
  - Hospital Pablo Tobon Uribe ( Site 0301), Medellín, Antioquia
  - Hospital General de Medellin Luz Castro de Gutierrez ( Site 0303), Medellín, Antioquia
  - Fundacion Valle del Lili ( Site 0300), Cali, Valle del Cauca Department
- General Hospital of Thessaloniki Hippokrateio ( Site 1402), Thessaloniki, Greece
- Norway (4):
  - Akershus Universitetssykehus HF ( Site 0903), Loerenskog, Akershus
  - Stavanger Universitetssykehus, Helse Stavanger ( Site 0901), Stavanger, Rogaland
  - St. Olavs Hospital ( Site 0900), Trondheim, Sor-Trondelag
  - Haukeland Universitetssjukehus ( Site 0902), Bergen, Vestfold
- Poland (2):
  - SPZOZ im. Dzieci Warszawy w Dziekanowie Lesnym ( Site 1002), Łomianki, Masovian Voivodeship
  - Wojewodzki Specjalistyczny Szpital im. Bieganskiego w Lodzi ( Site 1000), Lodz, Łódź Voivodeship
- Ukraine (6):
  - SI Dnipropetrovsk Regional Children Clinical Hospital DOR ( Site 1214), Dnipro, Dnipropetrovsk Oblast
  - Kharkiv City Children Hospital 16 ( Site 1200), Kharkiv, Kharkivs’ka Oblast’
  - Institution of Pediatr Obstetr and Gynec NAMS of Ukraine ( Site 1213), Kyiv, Kyivska Oblast
  - Odessa Regional Children Clinical Hospital ( Site 1203), Odesa, Odesa Oblast
  - Children City Clinical Hospital ( Site 1215), Poltava, Poltava Oblast
  - Zaporizhzhya Regional Clinical Childrens Hospital ( Site 1202), Zaporizhzhya, Zaporizhzhia Oblast
- United Kingdom (4):
  - Bristol Royal Hospital for Children ( Site 1101), Bristol, Bristol, City of
  - University Hospital Southampton NHS Foundation Trust ( Site 1100), Southampton, Hampshire
  - St. Georges University Hospital NHS Foundation Trust ( Site 1103), London, London, City of
  - Great Northern Children s Hospital ( Site 1102), Newcastle, Newcastle Upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Bradley JS, Makieieva N, Tondel C, Roilides E, Kelly MS, Patel M, Vaddady P, Maniar A, Zhang Y, Paschke A, Chen LF. Pharmacokinetics, Safety, and Tolerability of Imipenem/Cilastatin/Relebactam in Children with Confirmed or Suspected Gram-Negative Bacterial Infections: A Phase 1b, Open-Label, Single-Dose Clinical Trial. J Clin Pharmacol. 2023 Dec;63(12):1387-1397. doi: 10.1002/jcph.2334. Epub 2023 Sep 2. PMID 37562063

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note: Participant information is shown by age cohort and drug dosage to provide clinically-similar groups for analysis of participant baseline characteristics and safety data. Participant information in pharmacokinetic (PK) outcome measures is shown by age cohort, drug dose received and infusion time in order to provide appropriate and clinically discrete groups for PK analysis and modeling.
Groups:
- Cohort 1: IMI/REL 15/7.5 mg/kg: Adolescents (age 12 to <18 years) administered with a single intravenous (IV) 30-minute infusion dose of imipenem/cilastatin/relebactam (IMI/REL) at 15/7.5 mg/kg, up to maximum dose of 500/250 mg
- Cohort 2: IMI/REL 15/7.5 mg/kg: Older children (6 to <12 years) administered with a single IV 30-minute or 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg, up to a maximum dose of 500/250 mg
- Cohort 3: IMI/REL 15/7.5 mg/kg: Younger children (2 to <6 years) administered with a single IV 30-minute or 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg
- Cohort 4: IMI/REL 10/5 mg/kg: Infants (3 months to <1 year) administered with a single IV 60-minute infusion dose of IMI/REL at 10/5 mg/kg
- Cohort 4: IMI/REL 15/7.5 mg/kg: Toddlers (1 to <2 years) administered with a single IV 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg
- Cohort 5: Subcohort 1: IMI/REL 10/5 mg/kg: Young infants (4 weeks to <3 months of age) administered with a single IV 60-minute dose of IMI/REL at 10/5 mg/kg
- Cohort 5: Subcohort 2: IMI/REL 10/5 mg/kg: Older neonates (1 to <4 weeks of age) administered with a single IV 60-minute infusion dose of IMI/REL at 10/5 mg/kg
- Cohort 5: Subcohort 3: IMI/REL 10/5 mg/kg: Younger neonates (<1 week of age) administered with a single IV 60-minute infusion dose of IMI/REL at 10/5 mg/kg
- Cohort 5: Subcohort 1: IMI/REL 15/7.5 mg/kg: Young infants (4 weeks to <3 months of age) administered with a single IV 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg
- Cohort 5: Subcohort 2: IMI/REL 15/7.5 mg/kg: Older neonates (1 to <4 weeks of age) administered with a single IV 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg
- Cohort 5: Subcohort 3: IMI/REL 15/7.5 mg/kg: Younger neonates (<1 week of age) administered with a single IV 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg
Period: Overall Study
Arm/Group | Cohort 1: IMI/REL 15/7.5 mg/kg | Cohort 2: IMI/REL 15/7.5 mg/kg | Cohort 3: IMI/REL 15/7.5 mg/kg | Cohort 4: IMI/REL 10/5 mg/kg | Cohort 4: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 1: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 2: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 3: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 1: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 2: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 3: IMI/REL 15/7.5 mg/kg
Started | 7 | 6 | 6 | 4 | 4 | 6 | 3 | 2 | 2 | 3 | 4
Treated | 7 | 6 | 6 | 4 | 4 | 5 | 3 | 2 | 2 | 3 | 4
Completed | 7 | 6 | 6 | 4 | 4 | 5 | 3 | 2 | 2 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: IMI/REL 15/7.5 mg/kg | Cohort 2: IMI/REL 15/7.5 mg/kg | Cohort 3: IMI/REL 15/7.5 mg/kg | Cohort 4: IMI/REL 10/5 mg/kg | Cohort 4: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 1: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 2: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 3: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 1: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 2: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 3: IMI/REL 15/7.5 mg/kg | Total
Number analyzed (Participants) | 7 | 6 | 6 | 4 | 4 | 6 | 3 | 2 | 2 | 3 | 4 | 47
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 3 | 4 | 12
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 4 | 4 | 6 | 0 | 0 | 2 | 0 | 0 | 16
  Children (2-11 years) | 0 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12
  Adolescents (12-17 years) | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
  Adults (18-64 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 4 | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 28
  Male | 2 | 1 | 2 | 0 | 2 | 4 | 2 | 1 | 0 | 2 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 7
  Not Hispanic or Latino | 7 | 6 | 4 | 3 | 2 | 5 | 1 | 2 | 2 | 3 | 4 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 4
  White | 7 | 6 | 4 | 3 | 2 | 5 | 0 | 2 | 2 | 3 | 3 | 37
  More than one race | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Imipenem (IMI) Area Under the Concentration Time Curve From Time 0 to Infinity (AUC0-∞)
Description: Area under the concentration time curve from time 0 to infinity (AUC0-∞) of plasma imipenem (IMI) was calculated. AUC0-∞ is the area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time.
Time Frame: 30 minutes (min) before start of drug infusion (DI) and 10 min after the end of DI for all cohorts; 1.5 to 2.5 hours (hrs) and 4.5 to 6 hrs after start of DI for Cohorts 1-4; 2 to 5 hrs and 6 to 12 hrs after start of DI for Cohort 5
Population: All allocated participants who were compliant with the protocol and had at least 1 post-dose pharmacokinetic (PK) data point available for IMI AUC0-∞
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM*hr
Groups:
- Cohort 1: IMI/REL 500/250 mg 30-minute Infusion: Adolescents (age 12 to <18 years) administered with a single IV 30-minute infusion dose of IMI/REL at 500/250 mg
- Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion: Older children (6 to <12 years) administered with a single IV 30-minute infusion dose of IMI/REL at 15/7.5 mg/kg
- Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion: Older children (6 to <12 years) administered with a single IV 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg
- Cohort 2: IMI/REL 500/250 mg 30-minute Infusion: Older children (6 to <12 years) administered with a single IV 30-minute infusion dose of IMI/REL at 500/250 mg
- Cohort 2: IMI/REL 500/250 mg 60-minute Infusion: Older children (6 to <12 years) administered with a single IV 60-minute infusion dose of IMI/REL at 500/250 mg
- Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion: Younger children (2 to <6 years) administered with a single IV 30-minute infusion dose of IMI/REL at 15/7.5 mg/kg
- Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion: Younger children (2 to <6 years) administered with a single IV 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg
- Cohort 4: IMI/REL 10/5 mg/kg 60-minute Infusion: Infants (3 months to <1 year) administered with a single IV 60-minute infusion dose of IMI/REL at 10/5 mg/kg
- Cohort 4: IMI/REL 15/7.5 mg/kg 60-minute Infusion: Toddlers (1 to 2 years) administered with a single IV 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg
- Cohort 5: IMI/REL 10/5 mg/kg 60-minute Infusion: Neonates to infants (birth to <3 months of age) administered with a single IV 60-minute infusion dose of IMI/REL at 10/5 mg/kg
- Cohort 5: IMI/REL 15/7.5 mg/kg 60-minute Infusion: Neonates to infants (birth to <3 months of age) administered with a single IV 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 15/7.5 mg/kg 60-minute Infusion
Number analyzed (Participants) | 6 | 1 | 2 | 2 | 1 | 3 | 3 | 4 | 4 | 6 | 9
μM*hr | 134.7 (19.8) | 153.2 (NA) — NA=not calculated | 219.4 (39.2) | 139.4 (26.6) | 140 (NA) — NA=not calculated | 156 (18.9) | 163 (31.2) | 95.4 (39.3) | 219.2 (39.6) | 152.5 (14.1) | 271.3 (15.4)

2. Primary Outcome: IMI Maximum Concentration (Cmax)
Description: Maximum plasma concentration (Cmax) of IMI was calculated. Cmax is the peak plasma concentration of study drug after administration.
Time Frame: as for outcome 1
Population: All allocated participants who were compliant with the protocol and had at least 1 post-dose pharmacokinetic (PK) data point available for IMI Cmax
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 15/7.5 mg/kg 60-minute Infusion
Number analyzed (Participants) | 6 | 1 | 2 | 2 | 1 | 3 | 3 | 4 | 4 | 6 | 9
μM | 107.6 (16.4) | 126.0 (NA) — NA=not calculated | 123.0 (20.6) | 114.2 (9.2) | 110.6 (NA) — NA=not calculated | 150.3 (6.7) | 125.1 (25.2) | 64.9 (29.6) | 127.7 (36.0) | 79.4 (26.4) | 119.8 (16.8)

3. Primary Outcome: IMI Central Volume of Distribution (Vc)
Description: Central volume of distribution (Vc) of plasma IMI was calculated.
Time Frame: as for outcome 1
Population: All allocated participants who were compliant with the protocol and had at least 1 post-dose PK data point available for IMI Vc
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 15/7.5 mg/kg 60-minute Infusion
Number analyzed (Participants) | 6 | 1 | 2 | 2 | 1 | 3 | 3 | 4 | 4 | 6 | 9
Liters | 10.27 (16.2) | 8.00 (NA) — NA=not calculated | 4.33 (5.2) | 9.60 (2.4) | 8.70 (NA) — NA=not calculated | 3.49 (19.6) | 2.49 (34.6) | 2.39 (53.2) | 1.52 (35.0) | 1.06 (29.6) | 0.95 (34.2)

4. Primary Outcome: IMI Clearance (CL)
Description: Systemic clearance (CL) of plasma IMI was calculated.
Time Frame: as for outcome 1
Population: All allocated participants who were compliant with the protocol and had at least 1 post-dose PK data point available for IMI CL
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 15/7.5 mg/kg 60-minute Infusion
Number analyzed (Participants) | 6 | 1 | 2 | 2 | 1 | 3 | 3 | 4 | 4 | 6 | 9
L/hr | 12.58 (18.4) | 9.60 (NA) — NA=not calculated | 5.25 (9.2) | 11.67 (27.6) | 11.74 (NA) — NA=not calculated | 5.31 (29.7) | 4.43 (45.2) | 3.31 (60.1) | 1.70 (48.1) | 1.10 (26.2) | 0.66 (20.4)

5. Primary Outcome: IMI Percentage of Time Above the Minimum Concentration (%TMIC)
Description: Percentage of time spent above the minimum inhibitory concentration (%TMIC) of plasma IMI was calculated. %TMIC is defined as the percentage of time (in hours) in which the lowest concentration of a study drug, completely inhibits growth of the specific organism being tested.
Time Frame: as for outcome 1
Population: All allocated participants who were compliant with the protocol and had at least 1 post-dose PK data point available for IMI %TMIC
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of time
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 15/7.5 mg/kg 60-minute Infusion
Number analyzed (Participants) | 6 | 1 | 2 | 2 | 1 | 3 | 3 | 4 | 4 | 6 | 9
Percentage of time | 56.5 (17.1) | 58.3 (NA) — NA=not calculated | 80.3 (26.7) | 61.6 (25.1) | 56.7 (NA) — NA=not calculated | 50.1 (15.7) | 57.7 (18.8) | 50.4 (30.5) | 73.9 (19.7) | 70.2 (10.6) | 93.7 (9.3)

6. Primary Outcome: Relebactam (REL) AUC0-∞
Description: Area under the concentration time curve from time 0 to infinity (AUC0-∞) of plasma relebactam (REL) was calculated. AUC0-∞ is the area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time.
Time Frame: as for outcome 1
Population: All allocated participants who were compliant with the protocol and had at least 1 post-dose PK data point available for REL AUC0-∞
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM*hr
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 15/7.5 mg/kg 60-minute Infusion
Number analyzed (Participants) | 6 | 1 | 2 | 2 | 1 | 3 | 3 | 4 | 4 | 6 | 9
μM*hr | 80.1 (20.0) | 105.6 (NA) — NA=not calculated | 123.8 (59.5) | 90.3 (35.1) | 80.2 (NA) — NA=not calculated | 85.7 (32.4) | 81.7 (42.0) | 52.8 (33.6) | 126.6 (53.7) | 91.8 (18.3) | 220.7 (34.1)

7. Primary Outcome: REL Maximum Concentration (Cmax)
Description: Maximum plasma concentration (Cmax) of REL was calculated. Cmax is the peak plasma concentration of study drug after administration.
Time Frame: as for outcome 1
Population: All allocated participants who were compliant with the protocol and had at least 1 post-dose PK data point available for REL Cmax
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 15/7.5 mg/kg 60-minute Infusion
Number analyzed (Participants) | 6 | 1 | 2 | 2 | 1 | 3 | 3 | 4 | 4 | 6 | 9
μM | 49.33 (23.0) | 86.52 (NA) — NA=not calculated | 60.32 (30.7) | 57.44 (26.1) | 48.73 (NA) — NA=not calculated | 59.05 (9.08) | 48.59 (22.9) | 32.74 (15.0) | 59.55 (17.1) | 34.22 (17.3) | 61.04 (21.9)

8. Primary Outcome: REL Clearance (CL)
Description: Systemic clearance (CL) of plasma REL was calculated.
Time Frame: as for outcome 1
Population: All allocated participants who were compliant with the protocol and had at least 1 post-dose PK data point available for REL CL
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 15/7.5 mg/kg 60-minute Infusion
Number analyzed (Participants) | 6 | 1 | 2 | 2 | 1 | 3 | 3 | 4 | 4 | 6 | 9
L/hr | 8.98 (20.7) | 6.10 (NA) — NA=not calculated | 3.96 (28.9) | 8.03 (35.7) | 8.65 (NA) — NA=not calculated | 4.20 (40.8) | 3.65 (54.1) | 2.56 (54.5) | 1.27 (62.9) | 0.74 (27.0) | 0.35 (30.7)

9. Primary Outcome: REL Central Volume of Distribution (Vc)
Description: Central volume of distribution (Vc) of plasma REL was calculated.
Time Frame: as for outcome 1
Population: All allocated participants who were compliant with the protocol and had at least 1 post-dose PK data point available for REL Vc
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 10/5 mg/kg 60-minute Infusion | Cohort 5: IMI/REL 15/7.5 mg/kg 60-minute Infusion
Number analyzed (Participants) | 6 | 1 | 2 | 2 | 1 | 3 | 3 | 4 | 4 | 6 | 9
Liters | 10.58 (17.2) | 6.76 (NA) — NA=not calculated | 4.95 (1.6) | 9.81 (6.1) | 9.38 (NA) — NA=not calculated | 3.83 (13.8) | 2.88 (27.4) | 2.43 (38.8) | 1.70 (21.1) | 1.21 (24.6) | 0.90 (36.7)

10. Primary Outcome: Cilastatin (CIL) AUC0-∞
Description: Area under the concentration time curve from time 0 to infinity (AUC0-∞) of plasma cilastatin (CIL) was not calculated. AUC0-∞ is the area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time.
Time Frame: as for outcome 1
Population: Due to sparse PK sampling schedule, per participant data could not be calculated.
Groups:
- Cohort 1: IMI/REL 500-250 mg 30-minute Infusion: Cohort 1: IMI/REL 500/250 mg 30-minute infusion Adolescents (age 12 to <18 years) administered with a single IV 30-minute infusion dose of IMI/REL at 500/250 mg
- Cohort 4: IMI/REL 15/7.5 mg/kg: Toddlers (1 to 2 years) administered with a single IV 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg
- Cohort 5: IMI/REL 10/5 mg/kg: Neonates to infants (birth to <3 months of age) administered with a single IV 60-minute infusion dose of IMI/REL at 10/5 mg/kg
- Cohort 5: IMI/REL 15/7.5 mg/kg: Neonates to infants (birth to <3 months of age) administered with a single IV 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg
Arm/Group | Cohort 1: IMI/REL 500-250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg | Cohort 4: IMI/REL 15/7.5 mg/kg | Cohort 5: IMI/REL 10/5 mg/kg | Cohort 5: IMI/REL 15/7.5 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: CIL Time to Maximum Concentration (Tmax)
Description: Time to maximum plasma concentration (Tmax) of CIL was determined. Tmax is defined as the time after drug administration at which peak drug concentration in plasma occurs.
Time Frame: as for outcome 1
Population: All allocated participants who were compliant with the protocol and had at least 1 post-dose PK data point available for CIL Tmax
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg | Cohort 4: IMI/REL 15/7.5 mg/kg | Cohort 5: IMI/REL 10/5 mg/kg | Cohort 5: IMI/REL 15/7.5 mg/kg
Number analyzed (Participants) | 6 | 1 | 2 | 2 | 1 | 3 | 3 | 4 | 4 | 7 | 9
Hours | 0.58 [0.52 to 0.58] | 0.53 [0.53 to 0.53] | 1.1 [1.1 to 1.1] | 0.58 [0.57 to 0.58] | 1.1 [1.1 to 1.1] | 0.58 [0.57 to 0.58] | 1.1 [1.1 to 1.1] | 1.1 [1.1 to 1.7] | 1.2 [1.1 to 1.2] | 1.1 [1.1 to 1.2] | 1.2 [1.1 to 1.3]

12. Primary Outcome: CIL Concentration at End of Infusion (Ceoi)
Description: Concentration at end of infusion (Ceoi) of plasma CIL was determined.
Time Frame: 30 min after the start of infusion for Cohort 1; 60 min after the start of infusion for Cohorts 2-5
Population: All allocated participants who were compliant with the protocol and had at least 1 post-dose PK data point available for CIL Ceoi
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg | Cohort 4: IMI/REL 15/7.5 mg/kg | Cohort 5: IMI/REL 10/5 mg/kg | Cohort 5: IMI/REL 15/7.5 mg/kg
Number analyzed (Participants) | 6 | 1 | 2 | 2 | 1 | 3 | 3 | 3 | 4 | 7 | 9
μM | 86.9 (41.0) | 122 (NA) — Geometric coefficient of variation cannot be calculated for a sample size of 1. | 111 (51) | 80.5 (22) | 74.8 (NA) — Geometric coefficient of variation cannot be calculated for a sample size of 1. | 102 (32) | 80.9 (62) | 37.0 (64.0) | 94.5 (42.0) | 63.6 (28.0) | 107.0 (20.0)

13. Primary Outcome: CIL Terminal Half-Life (t1/2)
Description: Terminal half-life (t1/2) of plasma CIL was not calculated.
Time Frame: as for outcome 1
Population: Due to sparse PK sampling schedule, per participant data could not be calculated.
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg | Cohort 4: IMI/REL 15/7.5 mg/kg | Cohort 5: IMI/REL 10/5 mg/kg | Cohort 5: IMI/REL 15/7.5 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: CIL Clearance (CL)
Description: Systemic clearance (CL) of plasma CIL was not calculated.
Time Frame: as for outcome 1
Population: Due to sparse PK sampling schedule, per participant data could not be calculated.
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg | Cohort 4: IMI/REL 15/7.5 mg/kg | Cohort 5: IMI/REL 10/5 mg/kg | Cohort 5: IMI/REL 15/7.5 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: CIL Volume of Distribution (Vss)
Description: Volume of distribution (Vss) of plasma CIL was not calculated.
Time Frame: 30 minutes (min) before start of drug infusion (DI) and 10 min after the end of DI for all cohorts; 1.5 to 2.5 hours (hrs) and 4.5 to 6 hrs after start of DI for Cohorts 1-4; 2 to 5 hrs and 6 to12 hrs after start of DI for Cohort 5
Population: Due to sparse PK sampling schedule, per participant data could not be calculated.
Arm/Group | Cohort 1: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 2: IMI/REL 15/7.5 mg/kg mg 60-minute Infusion | Cohort 2: IMI/REL 500/250 mg 30-minute Infusion | Cohort 2: IMI/REL 500/250 mg 60-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 30-minute Infusion | Cohort 3: IMI/REL 15/7.5 mg/kg 60-minute Infusion | Cohort 4: IMI/REL 10/5 mg/kg | Cohort 4: IMI/REL 15/7.5 mg/kg | Cohort 5: IMI/REL 10/5 mg/kg | Cohort 5: IMI/REL 15/7.5 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: Number of participants with one or more AEs was calculated. An AE is defined as any untoward medical occurrence in a participant administered study drug and which may or may not have a causal relationship to the study drug.
Time Frame: Up to 17 days
Population: All allocated participants who received infusion (including partial doses) of study drug
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: IMI/REL 15/7.5 mg/kg: Adolescents (age 12 to <18 years) administered with a single IV 30-minute infusion dose of IMI/REL at 15/7.5 mg/kg, up to maximum dose of 500/250 mg
- Cohort 2: IMI/REL 15/7.5 mg/kg: Older children (6 to <12 years) administered with a single IV 30-minute or 60-minute infusion dose of IMI/REL at 15/7.5 mg/kg, up to maximum dose of 500/250 mg
Arm/Group | Cohort 1: IMI/REL 15/7.5 mg/kg | Cohort 2: IMI/REL 15/7.5 mg/kg | Cohort 3: IMI/REL 15/7.5 mg/kg | Cohort 4: IMI/REL 10/5 mg/kg | Cohort 4: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 1: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 2: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 3: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 1: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 2: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 3: IMI/REL 15/7.5 mg/kg
Number analyzed (Participants) | 7 | 6 | 6 | 4 | 4 | 5 | 3 | 2 | 2 | 3 | 4
Participants | 1 | 0 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: Number of participants who discontinued study drug due to an AE was calculated. An AE is defined as any untoward medical occurrence in a participant administered study drug and which may or may not have a causal relationship to the study drug.
Time Frame: Day 1
Population: All allocated participants who received infusion (including partial doses) of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: IMI/REL 15/7.5 mg/kg | Cohort 2: IMI/REL 15/7.5 mg/kg | Cohort 3: IMI/REL 15/7.5 mg/kg | Cohort 4: IMI/REL 10/5 mg/kg | Cohort 4: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 1: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 2: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 3: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 1: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 2: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 3: IMI/REL 15/7.5 mg/kg
Number analyzed (Participants) | 7 | 6 | 6 | 4 | 4 | 5 | 3 | 2 | 2 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 17 days (AE reporting), up to 19 days (all-cause mortality)
Description: The analysis population included all allocated participants who received infusion (including partial doses) of study drug. Note: Participant information is shown by age cohort and drug dosage, to provide clinically-similar groups for analysis of safety data.
Arm/Group | Cohort 1: IMI/REL 15/7.5 mg/kg | Cohort 2: IMI/REL 15/7.5 mg/kg | Cohort 3: IMI/REL 15/7.5 mg/kg | Cohort 4: IMI/REL 10/5 mg/kg | Cohort 4: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 1: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 2: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 3: IMI/REL 10/5 mg/kg | Cohort 5: Subcohort 1: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 2: IMI/REL 15/7.5 mg/kg | Cohort 5: Subcohort 3: IMI/REL 15/7.5 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/4 | 0/4 | 0/5 | 0/3 | 0/2 | 0/2 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/4 | 0/4 | 0/5 | 0/3 | 0/2 | 0/2 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 1/7 | 0/6 | 3/6 | 1/4 | 2/4 | 1/5 | 0/3 | 0/2 | 0/2 | 0/3 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: IMI/REL 15/7.5 mg/kg (N=7) | Cohort 2: IMI/REL 15/7.5 mg/kg (N=6) | Cohort 3: IMI/REL 15/7.5 mg/kg (N=6) | Cohort 4: IMI/REL 10/5 mg/kg (N=4) | Cohort 4: IMI/REL 15/7.5 mg/kg (N=4) | Cohort 5: Subcohort 1: IMI/REL 10/5 mg/kg (N=5) | Cohort 5: Subcohort 2: IMI/REL 10/5 mg/kg (N=3) | Cohort 5: Subcohort 3: IMI/REL 10/5 mg/kg (N=2) | Cohort 5: Subcohort 1: IMI/REL 15/7.5 mg/kg (N=2) | Cohort 5: Subcohort 2: IMI/REL 15/7.5 mg/kg (N=3) | Cohort 5: Subcohort 3: IMI/REL 15/7.5 mg/kg (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytoses (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT03230916/Prot_SAP_000.pdf